CLINICAL TRIAL: NCT01145833
Title: Guided Self-help Treatment for Families With an Overweight Child
Brief Title: Guided Self-help for Families With an Overweight Child
Acronym: GSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 081129; 1R21DK080266-01A1 (NIH)
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: obesity; guided self help treatment; treatment method; overweight; overweight children and parents; families with overweight child; efficacy; body mass index; weight
MeSH Terms: conditions — Obesity; Overweight; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate treatment group (Active Comparator): The immediate treatment group begins the 5-month treatment immediately after baseline assessment.
  Interventions: Other: Immediate Treatment Group
- Delayed Treatment Group (Other): The delayed treatment group serves as the control group. This group starts treatment 5 months after the baseline assessment. No intervention is involved during this 5-month waiting period. After 5 months, the delayed group is assessed for the second time and then begins the 5-month treatment.
  Interventions: Other: Delayed Treatment Group

INTERVENTIONS:
Other: Immediate Treatment Group — The immediate treatment group starts the 5-month treatment right after baseline assessment.
  Arms: Immediate treatment group
Other: Delayed Treatment Group — The delayed treatment group does not start treatment immediately after the baseline assessment. This group serves as the control group, by not receiving any treatment for 5 months. After the 5 months, the delayed group participants are asked to come in for a second assessment that involves completion of surveys and measurement of height, weight, and physical activity level. After this assessment is completed, the delayed group participants can begin the 5-month treatment.
  Other Names: Delayed Treatment Group (Control)
  Arms: Delayed Treatment Group

SUMMARY:
The purpose of this study is to evaluate whether a home based program can teach parents and moderately overweight kids who are of 8-12 years old with a BMI% between 85-97%, how to manage their child's weight. The study uses manuals and involves a short visit to the clinic every other week.

DETAILED DESCRIPTION:
An estimated 4-5 million children between the ages of 6-17 in the United States are obese. Children who are obese are at an increased risk for many negative health consequences in childhood and in adulthood. In addition, these children are at an increased risk for psychosocial consequences in childhood and adolescence, including poor self-esteem, teasing, verbal abuse and social isolation. Guided self-help offers an opportunity to provide empirically based programs to a larger amount of the target population. Once such treatment methods are available, it is possible that the guided self-help treatment for childhood obesity can be disseminated to primary care practitioners, psychologists, nurses, and health educators. Ultimately, the goal of this application is to develop a treatment protocol that can be used by clinics and lay health professionals to intervene with children who are overweight and their parents.

ELIGIBILITY:
Inclusion Criteria:

* child between the ages of 8 & 12
* an moderately overweight child with a BMI% between 85-97%
* child has a parent willing to participate
* child has a parent who can read English at a minimum of a 6th grade level
* family who is willing to commit to treatment attendance and attendance at all assessments.

Exclusion Criteria:

* Child psychiatric disorder diagnoses (based on parent report)
* Child diagnoses of a serious current physical disease (such as diabetes)
* Child who is taking medications that may impact their weight
* Child with physical difficulties that limit the ability to exercise
* Child with an active eating disorder
* Child and parent will be moving out of the San Diego County before study completion
* Child and/or parent has a modified diet due to religious or socially conscious reasons (such as Vegan, vegetarian)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD Center for Obesity and Health//Pediatrics Department, La Jolla, California, United States

REFERENCES:
- [Result] Epstein LH, Wing RR, Koeske R, Andrasik F, Ossip DJ. Child and parent weight loss in family-based behavior modification programs. J Consult Clin Psychol. 1981 Oct;49(5):674-85. doi: 10.1037//0022-006x.49.5.674. No abstract available. PMID 7287977
- [Result] Epstein LH, Kilanowski CK, Consalvi AR, Paluch RA. Reinforcing value of physical activity as a determinant of child activity level. Health Psychol. 1999 Nov;18(6):599-603. PMID 10619533
- [Result] Epstein LH, Myers MD, Raynor HA, Saelens BE. Treatment of pediatric obesity. Pediatrics. 1998 Mar;101(3 Pt 2):554-70. PMID 12224662
- [Result] Peterson CB, Mitchell JE, Engbloom S, Nugent S, Pederson Mussell M, Crow SJ, Thuras P. Self-help versus therapist-led group cognitive-behavioral treatment of binge eating disorder at follow-up. Int J Eat Disord. 2001 Dec;30(4):363-74. doi: 10.1002/eat.1098. PMID 11746298
- [Result] Epstein LH. Family-based behavioural intervention for obese children. Int J Obes Relat Metab Disord. 1996 Feb;20 Suppl 1:S14-21. PMID 8646260
- [Derived] Accurso EC, Norman GJ, Crow SJ, Rock CL, Boutelle KN. The role of motivation in family-based guided self-help treatment for pediatric obesity. Child Obes. 2014 Oct;10(5):392-9. doi: 10.1089/chi.2014.0023. Epub 2014 Sep 2. PMID 25181608
- [Derived] Boutelle KN, Norman GJ, Rock CL, Rhee KE, Crow SJ. Guided self-help for the treatment of pediatric obesity. Pediatrics. 2013 May;131(5):e1435-42. doi: 10.1542/peds.2012-2204. Epub 2013 Apr 1. PMID 23545372

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed Treatment Group: The delayed treatment group serves as the control group.
Period: Overall Study
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Started | 25 | 25
Completed | 22 | 25
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Delayed Treatment Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (1.3) | 10.5 (1.4) | 10.4 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 1 | 3
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Child BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (1.9) | 24.4 (2.6) | 24.2 (2.3)
Parent BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (6.1) | 27.9 (6.1) | 27.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Child BMI
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 22 | 25
kg/m^2 | 23.3 (2.1) | 25.17 (2.79)

2. Secondary Outcome: Parent BMI
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 22 | 25
kg/m^2 | 26.8 (6.4) | 28.0 (6.2)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No